CLINICAL TRIAL: NCT07162662
Title: Modulation of Gut Microbiota by Oral Sialic Acid: A Mechanistic Study
Brief Title: A Study on the Modulation of Gut Microbiota by Oral Sialic Acid in Healthy Subjects
Acronym: MFMOSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaolong Li (Other)
Responsible Party: Sponsor-Investigator, Xiaolong Li, Investigator, Army Medical University, China
Organization: Army Medical University, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-247-02; 2019R68 (Other Grant/Funding Number: ArmyMedChina); 2025-247-02 (Other: ArmyMedChina)
Record Dates: First submitted 2025-08-13; First posted 2025-09-09 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-09

CONDITIONS: Taking Sialic Acid to Regulate the Gut Microbiota; Healthy
Keywords: Oral Sialic Acid; Gut Microbiota; Healthy
MeSH Terms: interventions — N-Acetylneuraminic Acid

STUDY DESIGN:
Intervention Model Description: 1. Intervention: Oral administration of bird's nest peptide N-acetylneuraminic acid beverage produced by Huaxi Dankang Jiuhe Biotechnology Co., Ltd., with a daily dose of 500 mg (total 125ml) for 14 consecutive days.
  2. After volunteers are enrolled, fecal samples (5-7g) are collected before oral intervention. Immediately after collection, the fecal samples are stored at -80°C in the Department of General Surgery Laboratory for subsequent DNA extraction , gut microbiota analysis (16S rRNA sequencing) and Fecal Microbiota Transplantation (FMT) into mice (colorectal anastomosis model).
  3. Fourteen days after oral intervention, fecal samples (5-7g) are collected from the volunteers. Immediately after collection, the fecal samples are stored at -80°C in the Department of General Surgery Laboratory for subsequent DNA extraction, gut microbiota analysis (16S rRNA sequencing) and Fecal Microbiota Transplantation (FMT) into mice (colorectal anastomosis model).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- oral sialic acid (Experimental): This study employs a before-after self-control trial design, recruiting 42 volunteers to take oral sialic acid and collecting fecal samples before and after the intervention.
  Interventions: Dietary Supplement: Oral Sialic acid

INTERVENTIONS:
Dietary Supplement: Oral Sialic acid — This study employs a before-after self-control trial design, recruiting 42 volunteers to take oral sialic acid and collecting fecal samples before and after the intervention.

SUMMARY:
This is a single-center prospective cohort study conducted by the Department of General Surgery at the Second Affiliated Hospital of Army Medical University (Xinqiao Hospital). The purpose of this study is to explore and clarify the effects of sialic acid intervention on gut microbiota structure, with a focus on the proliferation of pathogens (e.g., Escherichia coli, Klebsiella pneumoniae), and to develop novel prevention and treatment strategies for improving intestinal homeostasis.

DETAILED DESCRIPTION:
Background：Colorectal cancer (CRC) is one of the most common gastrointestinal malignancies worldwide, ranking third in incidence and second in mortality among all cancers. Surgical resection remains the primary treatment for CRC, particularly for early- and mid-stage patients, as it effectively removes tumor tissue and prolongs survival. However, postoperative anastomotic healing failure (e.g., anastomotic leakage) is a severe complication of colorectal surgery, with an incidence rate of 5%-20%. Anastomotic leakage not only significantly increases postoperative mortality but also prolongs hospital stays, escalates medical costs, and imposes a heavy burden on both patients and healthcare systems. The pathogenesis of anastomotic leakage is complex, involving factors such as local ischemia, surgical technique, infection, and gut microbiota dysbiosis. In recent years, with advancements in microbiomics research, the role of gut microbiota in anastomotic healing has gained increasing attention.

During malignant transformation, colorectal cancer cells exhibit significantly upregulated expression of sialic acid (SA) on their cell surfaces. Sialic acid, a class of nine-carbon monosaccharides widely distributed on mammalian cell surfaces, participates in cell-cell recognition, immune regulation, and host-microbe interactions. Studies have shown that shed sialic acid from colorectal tumor cells enters the intestinal lumen, serving as a critical nutrient source for gut microbes. Notably, certain pathogens (e.g., Escherichia coli, Klebsiella pneumoniae) can utilize sialic acid as a carbon source to promote their proliferation and colonization. These pathogens may impair anastomotic healing through multiple mechanisms: first, by disrupting the intestinal mucosal barrier and exacerbating local inflammation; second, by inhibiting epithelial cell repair and delaying tissue regeneration; and third, by producing toxins or metabolites that further damage local tissues. Thus, colorectal tumor-derived sialic acid may indirectly increase the risk of postoperative anastomotic healing failure by nourishing specific pathogens.

Although existing research suggests that sialic acid from colorectal tumors influences the gut microenvironment by feeding pathogens, the specific mechanisms underlying its impact on postoperative anastomotic healing remain unclear. This hypothesis requires experimental validation. Our preliminary animal studies have demonstrated that oral administration of sialic acid impairs rectal anastomotic healing in mice by modulating gut microbiota. This finding indicates that sialic acid may affect postoperative anastomotic tissue repair and inflammatory responses by altering gut microbiota structure. However, research on the effects of sialic acid on the human gut microbiota remains limited. Based on this background, the present study aims to characterize the impact of sialic acid on gut microbiota by analyzing fecal samples collected from volunteers following oral sialic acid intervention.

Study Design： This study employs a before-after self-control trial design, recruiting 42 volunteers to take oral sialic acid and collecting fecal samples before and after the intervention. Specifically, the control group specimens were fecal samples collected before oral sialic acid administration, while the experimental group specimens were fecal samples collected after oral sialic acid administration.

Primary Objective:Alterations in Gut Microbiota Structure

Key Outcomes： Data Analysis: Data extracted from electronic medical records. Statistical analysis using SPSS 22.0 (χ² test for categorical data, t-test for normally distributed continuous data; significance p<0.05).

Ethics: Approved by the institutional ethics committee. Conducted in accordance with the Declaration of Helsinki and Chinese regulations. Patient privacy and data confidentiality are prioritized.

Timeline: Patient data collection and analysis (Sep 2025-Aug 2026); Statistical analysis and manuscript preparation (Sep-Dec 2025).

Significance:The purpose of this study is to explore and clarify the effects of sialic acid intervention on gut microbiota structure, with a focus on the proliferation of pathogens (e.g., Escherichia coli, Klebsiella pneumoniae), and to develop novel prevention and treatment strategies for improving intestinal homeostasis

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years
* No history of major diseases, no previous surgical history, and no history of cardiometabolic diseases (such as hypertension, diabetes mellitus, obesity, etc.)
* No use of drugs that may affect gut microbiota or metabolic function (e.g., antibiotics, probiotics, immunosuppressants, etc.);
* Voluntarily participate in the study and sign the informed consent form.

Exclusion Criteria:

* Comorbidities: Complicated with other severe diseases (e.g., immunodeficiency, chronic liver disease, renal insufficiency, malignant tumors, etc.).
* Recent infections: Registration records indicate a history of severe infections in the recent period (within 3 months) or currently receiving anti-infective treatment.
* Special populations: Pregnant women, lactating women, or women planning to become pregnant.
* Poor compliance: Volunteers who are unable to cooperate with the study protocol or follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Alterations in Gut Microbiota Structure | From enrollment to the end of treatment at 2 weeks
  Gut microbiota data analysis: Perform sequence analysis and OTU clustering using QIIME2 or Mothur; compare microbial diversity (α-diversity and β-diversity) between the experimental group and control group, as well as changes in the abundance of specific microbiota (e.g., Escherichia coli, Klebsiella pneumoniae); use LEfSe analysis to screen for microbiota with significant changes after sialic acid intervention, and predict changes in microbial functions via PICRUSt

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Army Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
We are currently planning to conduct a series of studies. As data sharing will be postponed until all studies have been completed, the data will not be made available at this time.